CLINICAL TRIAL: NCT03046355
Title: Timing of Delivery in Fetal Growth Restriction of Uncomplicated Women: A Randomized Controlled Trial (GROW Trial)
Brief Title: Timing of Delivery in Fetal Growth Restriction of Uncomplicated Women
Acronym: GROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Bahaeddine M Sibai, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-1053
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labor induction at 37.0 to 37.6 weeks of gestation (Experimental): Diagnosis of FGR with induction at 37 weeks 0 days of gestation to 37 weeks and 6 days
  Interventions: Procedure: Labor induction at 37.0 to 37.6 weeks of gestation
- Expectant monitoring until delivery (Active Comparator): Diagnosis of FGR managed with expectant monitoring and delivery as indicated
  Interventions: Procedure: Expectant monitoring until delivery

INTERVENTIONS:
Procedure: Labor induction at 37.0 to 37.6 weeks of gestation — Diagnosis of FGR with induction at 37 weeks 0 days of gestation to 37 weeks and 6 days
  Arms: Labor induction at 37.0 to 37.6 weeks of gestation
Procedure: Expectant monitoring until delivery — Diagnosis of FGR managed with expectant monitoring and delivery as indicated
  Arms: Expectant monitoring until delivery

SUMMARY:
The goal of the study is to determine whether labor induction at 37 weeks of pregnancy can improve the baby's health at birth when compared with delivery at a later point in the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age 34 weeks 0 days to 37 weeks 0 days at time of enrollment
* Dating of pregnancy by last menstrual period consistent with an ultrasound, ultrasound <21 weeks and 6 days of gestation, or known date of conception in the setting of in vitro fertilization
* No known major anomalies (anomalies requiring surgery antenatally or in the neonatal period, anomalies not compatible with life as determined by the physician)
* FGR defined as estimated fetal weight (EFW) < 10th percentile by Hadlock formula with normal umbilical artery Doppler studies and normal amniotic fluid

Exclusion Criteria:

* Known major fetal anomalies
* Multiple gestation or selective reduction of multiple gestation after 14 weeks
* Previous stillbirth at term
* Indications for delivery at <39 weeks. Common examples include:
* Placenta previa
* Placenta accreta
* Vasa previa
* History of classical cesarean section or myomectomy
* Human immunodeficiency virus (HIV)
* Oligohydramnios (low amniotic fluid, defined as maximum vertical pocket <2.0cm)
* High-risk pregnancy as determined by the physician. Common examples include:
* Pre-gestational diabetes or gestational diabetes on medication
* Chronic hypertension on medication
* Maternal cardiac disease
* Asthma requiring oral steroids during pregnancy
* Chronic renal disease
* Antiphospholipid syndrome
* Hyperthyroidism
* Prior stillbirth
* Systemic lupus erythematous
* Hemoglobinopathies such as sickle cell disease

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 21 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Number of children with birthweight less than the third percentile for gestational as assessed by NICHD nomograms | Immediately at birth
  NICHD is National Institute of Child Health and Human Development The NICHD nomogram will indicate their birth weight percentile based on their gestational age and ethnicity

SECONDARY OUTCOMES:
Number of children presenting with CNM | Up to 6 weeks after delivery
  Composite neo-natal morbidity (CNM) is any of the following: Apgar score <5 at 5 minutes, seizure, sepsis, hypoglycemia requiring intravenous treatment, mechanical ventilation, CPAP (continuous positive airway pressure) or high-flow nasal cannula for >2 hours, oxygen supplementation with FiO2 (fraction of inspired oxygen) >30% for >4 hours, death before discharge or IUFD (intrauterine fetal death).
Number of women presenting with CMM | Up to 6 weeks after delivery
  Composite maternal morbidity (CMM) is any of the following: chorioamnionitis, transfusion of blood products, endometritis, wound infection or separation, deep venous thrombosis, pulmonary embolism, admission to the intensive care unit, or death. Rates of cesarean section as well as indications in each group will also be evaluated.
Number of children delivered by cesarean section | Immediately at birth
Number of children admitted to NICU | Up to 6 weeks after delivery
  NICU is neo-natal intensive care unit
Number of children presenting with SGA | Immediately at birth
  SGA is small for gestational age when birthweight <10% for gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Baha M Sibai, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Bellaire - Memorial Hermann, Houston, Texas